CLINICAL TRIAL: NCT06751511
Title: The Effect of Inspiratory Muscle Warm-up on Decreased Diffusing Capacity for Carbon Monoxide After Maximal Exercise in Athletes: a Randomized, Placebo-controlled, Double-blind and Crossover Study
Brief Title: The Effect of Inspiratory Muscle Warm-up on Decreased Diffusing Capacity for Carbon Monoxide After Maximal Exercise in Athletes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emre Karaduman (Other)
Responsible Party: Sponsor-Investigator, Emre Karaduman, Research Asistant, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2023/473
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Athlete
Keywords: warm-up; inspiratory muscle warm-up; respiratory muscle warm-up

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Other): Participants only performed a general warm-up exercise.
  Interventions: Other: General warm-up
- IWM %15 Placebo (Placebo Comparator): In addition to the general warm-up, the participants performed IMW at 15% resistance intensity.
  Interventions: Other: Inspiratory muscle warm-up (Placebo - %15)
- IWM %40 Intervention (Active Comparator): In addition to the general warm-up, participants performed IMW at 40% resistance intensity.
  Interventions: Other: Inspiratory muscle warm-up (%40 IMW)

INTERVENTIONS:
Other: General warm-up — The General Warm-up (Control) protocol will consist of activities such as running and dynamic, active, and passive movements, adapted to suit the varied sports disciplines included in the study. These exercises will align with the principles of elevation, activation, and mobilization, aiming to enhance mobility across key muscle groups, from the arms and shoulders to the lower back and legs. Each session will include clear demonstrations to ensure proper technique and pacing, with participants performing a standardized number of repetitions. Researchers will supervise participants closely to verify accurate form and consistent execution during the intervention.
  Arms: Control
Other: Inspiratory muscle warm-up (Placebo - %15) — The placebo inspiratory muscle warm-up protocol will utilize the POWERbreathe® device at 15% of maximal inspiratory pressure (MIP). This placebo protocol will consist of two sets of 30 breaths, separated by a 60-second rest interval, with participants seated and wearing a nose clip. Proper technique will be taught during a prior familiarization session, and participants will be closely monitored during testing to ensure accurate execution. This protocol is designed to function as a placebo, effectively concealing the study's true objective to improve data validity and reliability.
  Arms: IWM %15 Placebo
Other: Inspiratory muscle warm-up (%40 IMW) — This study will implement a respiratory muscle warm-up protocol at 40% of maximal inspiratory pressure (MIP) using the POWERbreathe® device, as this intensity is considered optimal for effectively stimulating respiratory muscles. The protocol will consist of two sets of 30 breaths, with a 60-second rest period between sets, conducted while participants are seated and wearing a nose clip. Training for proper technique will be provided during the familiarization session, and participants will be closely monitored throughout the tests to ensure correct and consistent execution.
  Arms: IWM %40 Intervention

SUMMARY:
This study aims to examine the effects of inspiratory muscle warm-up (IMW) on the gas exchange capacity of the lungs (DLCO) and its potential contribution to recovery and athletic performance in elite athletes from various disciplines. The study hypothesizes that the decline in respiratory muscle capacity following high-intensity exercise, which negatively affects ventilation, diffusion, and oxygen transport, may be ameliorated through specific IMW protocol. A placebo-controlled, randomized, crossover, and double-blind design will be utilized, involving 28 elite male athletes from endurance, power, skill-based, and mixed disciplines.

Participants will complete three warm-up protocols: General Warm-up (GW), General Warm-up combined with IMW at 40% resistance intensity (GW+IMW40%), and a placebo condition (GW+IMWplacebo). Measurements will include respiratory muscle strength, DLCO (assessed at post-2, 30, 60, 90, and 120 minutes), respiratory function, and cardiorespiratory parameters during maximal exercise. This study is unique as it aims to detail the micro-level effects of IMW on pulmonary diffusion mechanisms and performance outcomes, providing novel insights into the ameliorative effects of IMW on respiratory function post-exercise. Additionally, it seeks to expand understanding of the mechanistic basis of IMW's benefits on both pulmonary diffusion capacity and athletic performance.

DETAILED DESCRIPTION:
STUDY DESIGN This study will employ a placebo-controlled, randomized, crossover, and double-blind research design to evaluate the effects of three warm-up conditions: Control, Placebo 15%, and IMW 40%. Athletes will be randomly assigned to the conditions using a crossover approach, ensuring that all participants will experience each protocol on separate days.

The warm-up protocols will include:

General Warm-up (Control): A standard warm-up without resistance. IMW 40%: A general warm-up combined with inspiratory muscle warm-up at 40% resistance intensity.

Placebo 15%: A general warm-up combined with inspiratory muscle warm-up (placebo) at 15% resistance intensity.

Blinding will be maintained for both participants and researchers. Participants will be informed that the study aims to investigate various warm-up types, while the true purpose will remain concealed. This design will ensure reliability and minimize bias in the data to be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-24 years.
* A training history of at least six years.
* Regular training frequency of at least four sessions per week.

Exclusion Criteria:

* History of smoking.
* History of physical disability or acute respiratory or cardiovascular disease within the past three months.
* Diagnosis of SARS-CoV-2 within the past three months.
* Pulmonary function measurements outside the normal clinical range (≤ 80%).

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Lung Carbon Monoxide Diffusion Capacity (DLCO) | Pre intervention and immediately post intervention
  DLCO will be measured using the single breath-hold method with a Quark PFT gas analyzer, following ATS/ERS standards. Each test involves inhalation of a gas mixture (0.3% CO, 0.3% CH4, and dry air), breath-holding for 10±2 seconds, and exhalation. Subjects will undergo DLCO tests at baseline, following the warm-up protocols, and at both the start and conclusion of VO2max testing. Additional measurements will be conducted at 2, 30, 60, 90, and 120 minutes post-VO2max during each laboratory visit.
Pulmonary Function (FVC) | Pre intervention and immediately post intervention
  Forced Vital Capacity (FVC) will be assessed using the Quark PFT device according to ATS/ERS guidelines. Subjects will perform the FVC maneuver while seated, with disposable mouthpieces and a nose clip to ensure accurate recordings. The FVC maneuver will involve a maximal inhalation followed by a rapid and forceful exhalation into the spirometer until no more air can be expelled. Subjects will be encouraged to maintain consistent effort throughout the maneuver to ensure reliable and reproducible results.
Pulmonary Function (SVC) | Pre intervention and immediately post intervention
  Slow Vital Capacity (SVC) will be assessed using the Quark PFT device according to ATS/ERS guidelines. Subjects will perform the SVC maneuver while seated, with disposable mouthpieces and a nose clip to ensure accurate recordings. The SVC maneuver will start with a full, deep inhalation. This will be followed by a slow and controlled exhalation at a steady pace until the lungs are completely emptied. The maneuver will provide measurements reflecting lung volumes under non-forced conditions.
Pulmonary Functions (MVV) | Pre intervention and immediately post intervention
  Maximum Voluntary Ventilation (MVV) will be assessed using the Quark PFT device according to ATS/ERS guidelines. Subjects will perform the MVV maneuver while seated, with disposable mouthpieces and a nose clip to ensure accurate recordings. The MVV maneuver will evaluate the maximum amount of air a subject can inhale and exhale in a specific timeframe, typically 12 seconds. Subjects will be instructed to breathe as quickly and deeply as possible during the maneuver. Proper coaching will be provided to help maintain maximal effort while avoiding hyperventilation-related discomfort.
Respiratory Muscle Strength | Pre intervention and immediately post intervention
  Respiratory muscle strength will be measured using the Pony FX MIP/MEP device following ERS guidelines. For maximal respiratory pressures, subjects will exhale maximally, followed by a maximal inspiration against a closed valve (and the opposite maneuver). At least three trials with less than 5% variability will be averaged to determine the final values.
Bicycle ergometer and Maximal Aerobic Capacity (VO2max) | Pre intervention and immediately post intervention
  The test will begin at a workload of 50 (Watt) and will progress by increasing the workload by 25 (Watt) every two minutes. Throughout the test, the pedaling speed (rhythm) will be continuously monitored on the bicycle display, and participants will be instructed to maintain a steady pace within an average range of ≥60 (±5) rpm. Despite strong verbal encouragement provided during the test, it will be terminated if a participant spends more than 10 seconds below the 55 rpm pedal rhythm and decides they cannot continue further (voluntary exhaustion). After completing the test, participants will continue pedaling at a workload of 20 (Watt) for approximately 2 minutes for active recovery. Each test will be initiated in accordance with the workload optimization and adjustments to bike fit (saddle, handlebar height, and position) performed during the first visit. Cardiopulmonary data will be obtained using a breath-by-breath Quark CPET metabolic system (Mixing chamber system) (COSMED).

IPD SHARING:
Plan to Share IPD: Undecided